CLINICAL TRIAL: NCT01982734
Title: Novel Strategies for the Enhancement of the Potency of Nutraceuticals With Low Oral Bioavailability and Their Application in Novel Functional Foods for Optimum Protection of the Aging Brain
Brief Title: Improved Oral Bioavailability of Curcumin Incorporated Into Micelles
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 051113-HS2
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Pharmacokinetics of New Curcumin Formulations; Safety of New Curcumin Formulations
Keywords: bioavailability; curcumin; pharmacokinetic; curcuma longa; age differences; sex differences
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Native curcumin (Active Comparator): 80 mg curcumin as native powder
  Interventions: Dietary Supplement: curcumin
- Native curcumin plus phytochemicals (Experimental): 80 mg curcumin as native powder plus 80 mg sesamin, 40 mg naringenin, 40 mg ferulic acid and 40 mg xanthohumol
  Interventions: Dietary Supplement: curcumin
- Curcumin micelles (Experimental): 80 mg curcumin incorporated into liquid micelles
  Interventions: Dietary Supplement: curcumin
- Curcumin micelles plus phytochemicals (Experimental): 80 mg curcumin incorporated into liquid micelles plus 80 mg sesamin, 40 mg naringenin, 40 mg ferulic acid, 40 mg xanthohumol incorporated into micelles
  Interventions: Dietary Supplement: curcumin

INTERVENTIONS:
Dietary Supplement: curcumin — 80 mg curcumin were given orally either as native powder, native powder plus phytochemicals,micelles or micelles plus phytochemicals

SUMMARY:
Curcumin, a lipophilic polyphenol derived from the plant curcuma longa possesses numerous health-promoting activities. The oral bioavailability of curcumin is low due to its poor aqueous solubility, limited gastrointestinal absorption, rapid metabolism and excretion. Therefore, we tested, in a randomized crossover study, simultaneous application of phytochemicals and micellar solubilisation, alone and together, as strategies to enhance the absorption of curcumin into the body. Furthermore, we investigated age and sex differences in curcumin pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with routine blood chemistry values within the normal ranges
* Age: 18-35 years or > 60 years

Exclusion Criteria:

* overweight (BMI >30 kg/m2)
* metabolic and endocrine diseases
* pregnancy
* lactation
* drug abuse
* use of dietary supplements or any form of medication (with the exception of oral contraceptives)
* smoking
* frequent alcohol consumption (>20 g ethanol/d)
* adherence to a restrictive dietary regimen
* physical activity of more than 5 h/wk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of total curcumin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Area under the plasma concentration versus time curve (AUC) of total demethoxycurcumin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Area under the plasma concentration versus time curve (AUC) of total bisdemethoxycurcumin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total curcumin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total demethoxycurcumin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total bisdemethoxycurcumin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total curcumin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total demethoxycurcumin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total bisdemethoxycurcumin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | 0, 4, 24h post-dose
Serum alanine transaminase activity [U/L] | 0, 4, 24h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 0, 4, 24h post-dose
Serum alkaline phosphatase activity [U/L] | 0, 4, 24h post-dose
Serum bilirubin [mg/dL] | 0, 4, 24h post-dose
Serum uric acid [mg/dL] | 0, 4, 24h post-dose
Serum creatinine [mg/dL] | 0, 4, 24h post-dose
Serum total cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum HDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum LDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum triacylglycerols [mg/dL] | 0, 4, 24h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Ph.D., Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Kocher, A., Schiborr, C., Behnam, D., & Frank, J. (2015). The oral bioavailability of curcuminoids in healthy humans is markedly enhanced by micellar solubilisation but not further improved by simultaneous ingestion of sesamin, ferulic acid, naringenin and xanthohumol. J Funct Foods 14: 183-19.
- See also: Website of the research group — http://www.nutrition-research.de/